CLINICAL TRIAL: NCT00880698
Title: Safety and Immunogenicity of a Live, Attenuated Rotavirus Vaccine (RotaTeq™) in HIV-1 Infected and Uninfected Children Born to HIV-1-Infected Mothers
Brief Title: Safety and Immune Response of a Rotavirus Vaccine in HIV-infected and Uninfected Children Born to HIV-infected Mothers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P1072; 10638 (Registry Identifier: DAIDS ES Registry ID); IMPAACT P1072
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Results first posted 2015-07-22 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2015-07

CONDITIONS: HIV Infection; Rotavirus Infection
Keywords: Rotavirus; Rotavirus vaccine
MeSH Terms: conditions — HIV Infections; Rotavirus Infections | interventions — RotaTeq

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HIV-uninfected RotaTeq (Experimental): HIV-1 uninfected participants receiving 3 doses of RotaTeq vaccine at intervals of 4-10 weeks with the third dose administered by 32 weeks of age.
  Interventions: Biological: RotaTeq
- HIV-uninfected Placebo (Placebo Comparator): HIV-1 uninfected participants receiving 3 doses of placebo at intervals of 4-10 weeks with the third dose administered by 32 weeks of age
  Interventions: Biological: Placebo
- HIV-infected RotaTeq (Experimental): HIV-1 infected participants receiving 3 doses of RotaTeq vaccine at intervals of 4-10 weeks with the third dose administered by 32 weeks of age.
  Interventions: Biological: RotaTeq
- HIV-1 infected Placebo (Placebo Comparator): HIV-1 infected participants receiving 3 doses of placebo at intervals of 4-10 weeks with the third dose administered by 32 weeks of age
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RotaTeq — 2 mL solution of live reassortant rotaviruses, containing G1, G2, G3, G4 and P1A which contains a minimum of 2.0 - 2.8 x 10^6 infectious units (IU) per individual reassortant dose, depending on the serotype, and not greater than 116 x 10^6 IUs per aggregate dose
  Arms: HIV-infected RotaTeq; HIV-uninfected RotaTeq
Biological: Placebo — 2 mL solution
  Arms: HIV-1 infected Placebo; HIV-uninfected Placebo

SUMMARY:
Rotavirus is the leading cause of severe diarrhea in infants and young children, accounting for 45% of severe diarrhea disease in both developed and developing countries. Annually, rotavirus causes approximately 111 million episodes of gastroenteritis requiring home care, 25 million clinic visits, 2 million hospitalizations, and approximately 440,000 deaths in children less than 5 years of age, of which approximately 90% of hospitalizations and 99% of deaths occur in developing countries. Although rotavirus infection is not more common in HIV-infected children, it complicates their care and interferes with their nutrition. Chances of death by these infections can be greater in HIV-infected children when they also suffer from wasting, malnutrition, and/or opportunistic infections. The primary purpose of this study was to evaluate the safety and immunogenicity of the Rotavirus vaccine candidate, RotaTeq, in HIV-infected and uninfected children born to HIV-infected mothers.

DETAILED DESCRIPTION:
International Maternal Pediatric Adolescent AIDS Clinical Trials Network (IMPAACT) P1072 was an international Phase II randomized double-blind study to assess the safety and immunogenicity of a live, attenuated rotavirus vaccine (RotaTeq) in HIV-1 infected (n=160) and uninfected (n=160) children born to HIV-1 infected mothers. Infants between 2 and <15 weeks of age at screening were assigned to one of four strata, based on HIV-1 status and in the HIV-1 infected, by Cluster of Differentiation percentage (CD4%) [≥ 20% (n=80), 15% ≤ CD4% < 20% (n=60) and < 15% (n=20)]. Screening had to be completed such that the first dose of study vaccine was administered when the participant was 4 to < 15 weeks of age. Within each stratum infants were randomized to receive either active RotaTeq vaccine (three doses of 2.0 mL each at intervals of 4 to 10 weeks with the third dose administered by 32 weeks of age) or placebo on the same schedule.

Participants were followed until six weeks after the last dose of vaccine, with visits at 7, 14, 21 and 42 days after each dose. The day 42 visit after the first two study doses was only required if the next study vaccination was done more than 42 days after the previous dose. At each visit, data were recorded on adverse events observed by the caretaker and investigator, including signs/symptoms ≥ grade 1 and new clinically significant diagnoses. No hematology or chemistry testing was required by the protocol, but sites could record laboratory results in the database if the results were pertinent. Stool samples for fecal shedding were collected at entry, days 7, 14, 21 and 42 after the first vaccination, 7 and 21 days after the second and third vaccinations, and at any unplanned visits for gastroenteritis. Serum for immunogenicity testing was collected at entry and 14 days (or 42 days if not collected at 14 days) after the third vaccination.

In January 2012, rotavirus vaccine (Rotarix) became available as standard of care at the Lusaka study site in Zambia, so enrollment ceased at that site. Infants already enrolled and within the age range where they could receive the Rotarix series were unblinded. Those on placebo were given Rotarix. Those in the active vaccine arm continued receiving the study vaccine. All infants continued to attend study visits. A similar procedure was followed after July 2012, when Rotarix became available as standard of care in Botswana.

During 2013, Zimbabwe was the only site enrolling participants, most of whom were HIV-1 uninfected. The team decided to close the study to enrollment prematurely at the end of September 2013 with a total of 126 HIV-1 uninfected (79% of the target of 160) and 76 HIV-1 infected (48% of the target: 81% of those with CD4% ≥ 20% and 14% of those with CD4% < 20%). Because of the low enrollment of HIV-1 infected infants with lower CD4%, results in the HIV-1 infected stratum were reported combined across CD4% strata.

Baseline characteristics are presented 'as-randomized'. Safety data are presented 'as-randomized' and include all follow-up on study up to 42 days after the third vaccination. Immunogenicity results are presented for the 'per-protocol' population which includes participants who received the 'as-randomized' vaccine and completed the three vaccinations within the required windows (first vaccination between 4 and < 15 weeks of age, subsequent vaccinations at least 28 days after previous vaccination, and third dose by 32 weeks of age).

ELIGIBILITY:
Inclusion Criteria for All Vaccinations:

* Participant was born to an HIV-1-infected mother whose HIV-1 diagnosis was determined by two different tests performed on the same or separate maternal samples obtained before or during pregnancy or during the post-partum period. Acceptable tests are antibodies in serum or saliva, HIV RNA or DNA, or antigen in the blood.
* Presence or absence of HIV RNA or DNA in the blood of the infant
* CD4% documented at screening
* Parent or legal guardian agreed to give written informed consent and was willing to comply with study requirements
* Parents/guardians of each participant stated their willingness to have the child follow the country-specific childhood Expanded Programme on Immunization ("EPI") schedule for concomitant childhood vaccines recommended during the study period
* HIV-infected participants had initiated antiretroviral therapy (ART) before or at the time of administration of the first dose of study vaccine/placebo. Note: It was not acceptable for participants to take a prescription home with them to start ART on the day of vaccination.

Inclusion Criteria for second and third vaccinations:

* Successful administration of first vaccine (for second vaccination) and second vaccine (for third vaccination)
* Participants were less than 32 weeks of age at the time of the third vaccine/placebo dose

Exclusion Criteria for All Vaccinations:

* Concurrent participation in any study of an investigational drug or vaccine, except for studies for prevention of perinatal HIV-1 transmission
* Known allergy to any component of the study vaccine
* Active gastrointestinal illness or fever. Fever was defined as greater than or equal to 38.5º C in accordance with WHO guidelines for administration of childhood vaccines.
* Could not be enrolled from any site at which rotavirus vaccine was available and was being administered
* Any condition, which would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol
* Any other condition, situation, or clinically significant finding (other than HIV infection) that, in the investigator's opinion, would interfere with study participation, or interpretation
* Participants with a known history of Severe Combined Immunodeficiency (SCID) or intussusception

Exclusion Criteria for second and third vaccinations:

- Any Grade 4 adverse events believed to be possibly/probably/definitely related to vaccine would disqualify subjects from receiving additional doses. Grade 3 adverse events believed to be possibly/probably related to vaccine had to be demonstrated to have improved to less than Grade 2 prior to receiving the next scheduled dose.

Ages: 2 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2009-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron J. Levin, MD, Study Chair — University of Colorado at Denver Health Sciences Center
Locations (6):
- Botswana (2):
  - Gaborone CRS, Gaborone
  - Molepolole CRS, Gaborone
- Kilimanjaro Christian Medical Center CRS, Moshi, Tanzania
- George CRS, Lusaka, Zambia
- Zimbabwe (2):
  - Harare Family Care CRS, Harare
  - Parirenyatwa CRS, Harare

REFERENCES:
- [Background] Committee on Infectious Diseases; American Academy of Pediatrics. Prevention of rotavirus disease: updated guidelines for use of rotavirus vaccine. Pediatrics. 2009 May;123(5):1412-20. doi: 10.1542/peds.2009-0466. Epub 2009 Mar 30. PMID 19332437
- [Background] Kiulia NM, Nyaundi JK, Peenze I, Nyachieo A, Musoke RN, Steele AD, Mwenda JM. Rotavirus infections among HIV-infected children in Nairobi, Kenya. J Trop Pediatr. 2009 Oct;55(5):318-23. doi: 10.1093/tropej/fmp016. Epub 2009 Mar 10. PMID 19276145
- [Background] Parashar UD, Glass RI. Rotavirus vaccines--early success, remaining questions. N Engl J Med. 2009 Mar 12;360(11):1063-5. doi: 10.1056/NEJMp0810154. No abstract available. PMID 19279338
- [Derived] Levin MJ, Lindsey JC, Kaplan SS, Schimana W, Lawrence J, McNeal MM, Bwakura-Dangarembizi M, Ogwu A, Mpabalwani EM, Sato P, Siberry G, Nelson M, Hille D, Weinberg GA, Weinberg A. Safety and immunogenicity of a live attenuated pentavalent rotavirus vaccine in HIV-exposed infants with or without HIV infection in Africa. AIDS. 2017 Jan 2;31(1):49-59. doi: 10.1097/QAD.0000000000001258. PMID 27662551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at five sites in four sub-saharan countries: Botswana (2), Tanzania, Zambia and Zimbabwe between December 2009 and October 2013.
Pre-assignment Details: Enrollment of infants 2 to < 15 weeks of age was stratified by HIV-1 infection and within the HIV-1 infected stratum, by CD4% (<15%, 15%-<20% and >=20%). Within stratum, participants were randomized with equal probability to receive three doses of RotaTeq or Placebo.
Period: Overall Study
Arm/Group | HIV-uninfected RotaTeq | HIV-uninfected Placebo | HIV-infected RotaTeq | HIV-1 Infected Placebo
Started | 62 | 64 | 37 | 39
Completed | 61 | 61 | 36 | 36
Not Completed | 1 | 3 | 1 | 3
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes all participants 'as randomized'
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-uninfected RotaTeq | HIV-uninfected Placebo | HIV-infected RotaTeq | HIV-1 Infected Placebo | Total
Number analyzed (Participants) | 62 | 64 | 37 | 39 | 202
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 82 [71 to 92] | 79 [71 to 92] | 92 [82 to 94] | 93 [83 to 99] | 87 [75 to 94]
Age, Customized [Number; unit: Participants]
  27-42 days | 5 | 2 | 1 | 0 | 8
  43-84 days | 29 | 39 | 10 | 10 | 88
  85-105 days | 28 | 23 | 26 | 29 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 19 | 22 | 108
  Male | 29 | 30 | 18 | 17 | 94
Region of Enrollment [Number; unit: participants]
  Botswana | 19 | 18 | 17 | 16 | 70
  Tanzania | 3 | 4 | 2 | 4 | 13
  Zimbabwe | 36 | 38 | 16 | 15 | 105
  Zambia | 4 | 4 | 2 | 4 | 14
Ever breast fed [Number; unit: participants]
  Yes | 36 | 43 | 22 | 26 | 127
  No | 26 | 21 | 15 | 13 | 75
Screening CD4 percent (%) [Median (Inter-Quartile Range); unit: percent] | 37 [33 to 45] | 38 [31 to 45] | 31 [24 to 38] | 29 [23 to 34] | 35 [28 to 43]
HIV-1 RNA (copies/ml) [Median (Inter-Quartile Range); unit: copies/ml] — HIV-1 RNA not collected in HIV-1 uninfected stratum. HIV-1 infected RotaTeq (n=35), Placebo (n=37). Upper limit of detection of HIV-1 RNA assay is 750,000 copies/ml.
  copies/ml | NA [NA to NA] — Not collected in HIV-1 uninfected cohort | NA [NA to NA] — Not collected in HIV-1 uninfected cohort | 39827 [1380 to 569000] | 83628 [9660 to 750000] | NA [NA to NA] — Not collected in HIV-1 uninfected cohort

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Developing New Grade >=3 Adverse Events
Description: Percentage of participants developing new grade >=3 adverse events (abnormal laboratory values (hematology and chemistry), signs, symptoms and diagnoses) not present at the time of the first vaccination. Adverse events were graded using the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (Version 1.0, December 2004, Clarification August 2009).
Time Frame: From study entry until at least 42 days after third vaccination
Population: Participants classified 'as'randomized'. Includes all follow-up on participants unblinded during the study and found to be on RotaTeq. Follow-up on participants unblinded during the study and found to be on placebo censored at the time of their last study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HIV-uninfected RotaTeq | HIV-uninfected Placebo | HIV-infected RotaTeq | HIV-1 Infected Placebo
Number analyzed (Participants) | 62 | 64 | 37 | 39
Percentage of participants | 1.6 [0.0 to 8.7] | 4.7 [1.0 to 13.1] | 13.5 [4.5 to 28.8] | 12.8 [4.3 to 27.4]
Statistical Analysis 1: Comparison: HIV-uninfected RotaTeq vs HIV-uninfected Placebo; Test type: Superiority or Other; p = 0.62, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = -3.1, 95% CI 2-sided [-20.6 to 14.8] — Difference and 95% confidence interval (RotaTeq minus Placebo) in percentage of HIV-uninfected participants experiencing a new grade >=3 adverse event
Statistical Analysis 2: Comparison: HIV-infected RotaTeq vs HIV-1 Infected Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 0.7, 95% CI 2-sided [-21.0 to 23.4] — Difference and 95% confidence interval (RotaTeq minus Placebo) in percentage of HIV-infected participants experiencing a new grade >=3 adverse event

2. Primary Outcome: Percentage of Participants Classified as Responders as Measured by Serum Anti-rotavirus IgA ELISA (IgA) and Serum Neutralizing Antibodies (SNA) G1, G2, G3, G4 and P1.
Description: Percentage of participants who experienced >=3-fold increases from prior to the first vaccination to at least 14 days after the third vaccination in Iga, SNA G1, SNA G2, SNA G3, SNA G4 and SNA P1.
Time Frame: Prior to first vaccination and at least 14 days after third vaccination
Population: Only participants in the per-protocol population (received all 3 as-randomized vaccinations within recommended windows) and with measurements prior to the first vaccination and at least 11 days after the third vaccination and whose levels at the entry time point were less than one third of the upper limit of detection of the assay were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HIV-uninfected RotaTeq | HIV-uninfected Placebo | HIV-infected RotaTeq | HIV-1 Infected Placebo
Number analyzed (Participants) | 57 | 58 | 34 | 32
Percentage of participants
  SNA G1 | 31.6 [19.9 to 45.2] | 1.7 [0.0 to 9.2] | 52.9 [35.1 to 70.2] | 3.1 [0.1 to 16.2]
  SNA G2 | 12.3 [5.1 to 23.7] | 5.2 [1.1 to 14.4] | 23.5 [10.7 to 41.2] | 9.4 [2.0 to 25.0]
  SNA G3 | 21.1 [11.4 to 33.9] | 1.7 [0.0 to 9.2] | 29.4 [15.1 to 47.5] | 0.0 [0.0 to 10.9]
  SNA G4 | 31.6 [19.9 to 45.2] | 5.2 [1.1 to 14.4] | 61.8 [43.6 to 77.8] | 3.1 [0.1 to 16.2]
  SNA P1 (Uninfect Rot n=56; Infect Rot n=33) | 25.0 [14.4 to 38.4] | 8.6 [2.9 to 19.0] | 24.2 [11.1 to 42.3] | 12.5 [3.5 to 29.0]
  IgA (Infect RotaTeq n=32; Placebo n=31) | 80.7 [68.1 to 90.0] | 29.3 [18.1 to 42.7] | 81.3 [63.6 to 92.8] | 16.1 [5.5 to 33.7]
Statistical Analysis 1: Comparison: HIV-uninfected RotaTeq vs HIV-uninfected Placebo; SNA G1; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 29.9, 95% CI 2-sided [11.5 to 46.1] — Difference (95% confidence interval) in percentage of HIV-1 uninfected participants classified as responders for SNA G1 in RotaTeq group minus Placebo group
Statistical Analysis 2: Comparison: HIV-infected RotaTeq vs HIV-1 Infected Placebo; SNA G1; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 49.8, 95% CI 2-sided [27.1 to 68.6] — Difference (95% confidence interval) in percentage of HIV-1 infected participants classified as responders for SNA G1 in RotaTeq group minus Placebo group
Statistical Analysis 3: Comparison: HIV-uninfected RotaTeq vs HIV-uninfected Placebo; SNA G2; Test type: Superiority or Other; p = 0.20, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 7.1, 95% CI 2-sided [-11.3 to 24.8] — Difference (95% confidence interval) in percentage of HIV-1 uninfected participants classified as responders for SNA G2 in RotaTeq group minus Placebo group
Statistical Analysis 4: Comparison: HIV-infected RotaTeq vs HIV-1 Infected Placebo; SNA G2; Test type: Superiority or Other; p = 0.19, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 14.2, 95% CI 2-sided [-10.6 to 36.7] — Difference (95% confidence interval) in percentage of HIV-1 infected participants classified as responders for SNA G2 in RotaTeq group minus Placebo group
Statistical Analysis 5: Comparison: HIV-uninfected RotaTeq vs HIV-uninfected Placebo; SNA G3; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 19.3, 95% CI 2-sided [0.9 to 36.4] — Difference (95% confidence interval) in percentage of HIV-1 uninfected participants classified as responders for SNA G3 in RotaTeq group minus Placebo group
Statistical Analysis 6: Comparison: HIV-infected RotaTeq vs HIV-1 Infected Placebo; SNA G3; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 29.4, 95% CI 2-sided [4.7 to 50.6] — Difference (95% confidence interval) in percentage of HIV-1 infected participants classified as responders for SNA G3 in RotaTeq group minus Placebo group
Statistical Analysis 7: Comparison: HIV-uninfected RotaTeq vs HIV-uninfected Placebo; SNA G4; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 26.4, 95% CI 2-sided [8.0 to 42.9] — Difference (95% confidence interval) in percentage of HIV-1 uninfected participants classified as responders for SNA G4 in RotaTeq group minus Placebo group
Statistical Analysis 8: Comparison: HIV-infected RotaTeq vs HIV-1 Infected Placebo; SNA G4; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 58.6, 95% CI 2-sided [37.2 to 75.9] — Difference (95% confidence interval) in percentage of HIV-1 infected participants classified as responders for SNA G4 in RotaTeq group minus Placebo group
Statistical Analysis 9: Comparison: HIV-uninfected RotaTeq vs HIV-uninfected Placebo; SNA P1; Test type: Superiority or Other; p = 0.024, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 16.4, 95% CI 2-sided [-1.7 to 34.2] — Difference (95% confidence interval) in percentage of HIV-1 uninfected participants classified as responders for SNA P1 in RotaTeq group minus Placebo group
Statistical Analysis 10: Comparison: HIV-infected RotaTeq vs HIV-1 Infected Placebo; SNA P1; Test type: Superiority or Other; p = 0.34, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 11.7, 95% CI 2-sided [-12.0 to 35.5] — Difference (95% confidence interval) in percentage of HIV-1 infected participants classified as responders for SNA P1 in RotaTeq group minus Placebo group
Statistical Analysis 11: Comparison: HIV-uninfected RotaTeq vs HIV-uninfected Placebo; IgA; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 51.4, 95% CI 2-sided [34.3 to 66.3] — Difference (95% confidence interval) in percentage of HIV-1 uninfected participants classified as responders for IgA in RotaTeq group minus Placebo group
Statistical Analysis 12: Comparison: HIV-infected RotaTeq vs HIV-1 Infected Placebo; IgA; Test type: Superiority or Other; p < 0.001, Fisher Exact — The pre-specified significance level was 5%. No adjustments were made for multiple comparisons; Risk Difference (RD) = 65.1, 95% CI 2-sided [42.7 to 81.7] — Difference (95% confidence interval) in percentage of HIV-1 infected participants classified as responders for IgA in RotaTeq group minus Placebo group

3. Secondary Outcome: Number of Participants With Fecal Shedding of RotaTeq Strains After Each Vaccination
Description: Number of participants with at least one positive enzyme immuno assay (EIA) rotavirus antigen test, positive fluorescent focal assay, and specific for rotavirus gene 6 which codes for the VP6 protein after each vaccination.
Time Frame: At entry, days 7, 14, 21 and 42 days after first dose, and at days 7 and 21 after the second and third doses
Population: All participants 'as randomized'
Measure: Number; unit: participants
Arm/Group | HIV-uninfected RotaTeq | HIV-uninfected Placebo | HIV-infected RotaTeq | HIV-1 Infected Placebo
Number analyzed (Participants) | 62 | 64 | 37 | 39
participants
  Post dose 1 | 0 | 0 | 1 | 0
  Post dose 2 | 0 | 0 | 0 | 0
  Post dose 3 | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of HIV-1 Infected Participants With HIV-1 RNA <= 400 Copies/ml
Description: Percentage of HIV-1 infected participants with HIV-1 RNA <= 400 copies/ml at last study visit
Time Frame: 42 days after third vaccination or last study visit with an HIV-1 RNA measurement
Population: Includes HIV-infected participants 'as-randomized' with an HIV-1 RNA measurement at their last study visit
Measure: Number; unit: Percentage of participants
Arm/Group | HIV-infected RotaTeq | HIV-1 Infected Placebo
Number analyzed (Participants) | 35 | 34
Percentage of participants | 54.3 | 44.1

5. Secondary Outcome: Change in CD4 Percent From Entry to Last Study Visit in HIV-1 Infected Participants
Description: Change calculated as value at last study visit minus value closest to and before randomization date
Time Frame: At entry and 42 days after third vaccination or last study visit with CD4 measurement
Population: Includes HIV-1 infected participants 'as-randomized' with a CD4 percent measurement prior to first vaccination and at last study visit
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | HIV-infected RotaTeq | HIV-1 Infected Placebo
Number analyzed (Participants) | 36 | 35
Percentage of lymphocytes | 3 (7.0) | 3 (8.7)

6. Secondary Outcome: Change in CD4 Count From Entry to Last Study Visit in HIV-1 Infected Participants
Description: Change calculated as value at last study visit minus value closest to and before randomization date
Time Frame: At entry and 42 days after third vaccination or last study visit with CD4 measurement
Population: Includes HIV-infected participants 'as randomized' with a CD4 count measurement prior to first vaccination and at their last study visit
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | HIV-infected RotaTeq | HIV-1 Infected Placebo
Number analyzed (Participants) | 36 | 35
cells/mm^3 | 201 (1060) | 335 (1031)

7. Secondary Outcome: Number of Participants Classified at Screening or Entry as HIV-1 Uninfected, and Acquiring HIV-1 Infection on Study
Description: HIV tests were done at screening, entry and the last study visit after the third vaccination. Any participants classified as HIV-1 uninfected at screening or entry but HIV-1 infected at their last study visit would be classified as acquiring HIV-1 infection during the study
Time Frame: From study entry until at least 42 days after third vaccination
Population: Includes HIV-1 uninfected participants 'as-randomized' with an HIV test at entry and either 2 or 6 weeks after the third vaccination (or after the time point at which they would have received the third vaccination if they did not receive all three doses)
Measure: Number; unit: participants
Arm/Group | HIV-uninfected RotaTeq | HIV-uninfected Placebo
Number analyzed (Participants) | 61 | 60
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From study enrollment until study completion (up to 24 weeks)
Description: The Serious Adverse Event (SAE) reporting category defined in V2.0 of the Division of AIDS (DAIDS) Expedited (EAE) Manual was used in addition to all cancers and vaccine overdoses. AEs were graded using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, V1.0, Dec. 2004.
Arm/Group | HIV-1 Uninfected RotaTeq | HIV-1 Uninfected Placebo | HIV-1 Infected RotaTeq | HIV-1 Infected Placebo
Serious Adverse Events (participants affected / at risk) | 2/62 | 4/64 | 5/37 | 4/39
Other Adverse Events (participants affected / at risk) | 39/62 | 39/64 | 29/37 | 29/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-1 Uninfected RotaTeq (N=62) | HIV-1 Uninfected Placebo (N=64) | HIV-1 Infected RotaTeq (N=37) | HIV-1 Infected Placebo (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 1
Malaria (Infections and infestations) | 0 | 1 | 0 | 0
Measles (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-1 Uninfected RotaTeq (N=62) | HIV-1 Uninfected Placebo (N=64) | HIV-1 Infected RotaTeq (N=37) | HIV-1 Infected Placebo (N=39)
Otorrhoea (Ear and labyrinth disorders) | 5 | 0 | 0 | 1
Conjunctival pallor (Eye disorders) | 0 | 1 | 2 | 0
Eye discharge (Eye disorders) | 3 | 5 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 19 | 15 | 14 | 10
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 8 | 10 | 10 | 6
Feeling hot (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 16 | 12 | 11 | 15
Conjunctivitis (Infections and infestations) | 3 | 4 | 1 | 0
Gastroenteritis (Infections and infestations) | 9 | 6 | 4 | 3
Oral candidiasis (Infections and infestations) | 2 | 1 | 1 | 4
Otitis media (Infections and infestations) | 4 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 3 | 0
Haemoglobin decreased (Investigations) | 0 | 3 | 2 | 3
Neutrophil count decreased (Investigations) | 0 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 25 | 20 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 8 | 10
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 | 12 | 8 | 10
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 5 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 6
Eczema infantile (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 10 | 11 | 10 | 10
Rash generalised (Skin and subcutaneous tissue disorders) | 3 | 8 | 5 | 7
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
The study was closed to enrollment prematurely so statistical power to detect differences was reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.